CLINICAL TRIAL: NCT04852614
Title: Pharmacokinetics of Sofosbuvir/Daclatasvir in HCV-infected Lactating Women: a Pilot Study
Brief Title: Pharmacokinetics of Sofosbuvir/Daclatasvir in HCV-infected Lactating Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manal Hamdy El-Sayed, Director of Faculty of Medicine Ain Shams University Research Institute, Ain Shams University
Other Study IDs: CL 2489
Record Dates: First submitted 2021-04-17; First posted 2021-04-21 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Hepatitis C Virus Infection
Keywords: Egypt; Sofosbuvir/daclatasvir; Pharmacokinetics; Lactating Women
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pharmacokinetic test — Blood samples will be collected 48 hours after the first dose on day 3 of the observed intake of the study medication at the following time points: t=0 (pre-dose), 1, 2, 3, 4, 8 and 12 hours post ingestion (7 samples) (3 mL each), Breast milk samples will be collected by emptying both breasts at 0, 2, 4, 8 and 12 hours (5 samples).

SUMMARY:
This is a prospective, observational, open-label, pharmacokinetic study will evaluate PK of SOF/DAC in lactating HCV-infected females at weaning or women who voluntarily decided to forego breastfeeding to initiate HCV infection treatment. Therefore, drug concentrations can be determined in maternal plasma and milk without risk to the children. HCV infected women at weaning after various durations of breastfeeding and HCV infected women who wish to initiate treatment immediately after delivery and forego breastfeeding will be recruited to start treatment under the guidance of their physician with SOF/DAC to determine M/P ratios of each of SOF, GS-331007 and DAC.

DETAILED DESCRIPTION:
Eligible women will be advised to arrange for initiation of treatment with their physician once they decide to stop breastfeeding. Treatment will be initiated once the women decide to wean their children and a warning will be given to abstain from any breast-feeding once treatment is started. This treatment is prescribed by the physician either the patients choose to participate in the study or not. In addition, effective contraceptive methods should be used. The treatment consists of SOF/DAC: 400 mg sofosbuvir and 60 mg daclatasvir administered with food for 12 weeks.

All recruited patients will be screened for the following data at baseline: Serum creatinine, bilirubin, albumin, AST, ALT, prothrombin time (PT), CBC, and viral load by PCR. The patient's general and demographic information (age, gender, height, and weight), comorbidities, and concurrent medications will be assessed and recorded in a specially designed patient data sheet.

The study will be conducted in the Faculty of Medicine Ain-Shams Research Institute Clinical Research Center (MASRI -CRC). After the first dose, women will be instructed to express their milk and discard it on the first two days and come to the research center on the third day for plasma and milk sampling. Patients will be instructed to take the dose on time especially the day before sampling. They will be asked to record the time of dose administration. They might be also followed up by telephone calls

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age at the day of screening.
* Confirmed HCV infection by PCR and known genotype (GT) 1, 4, 5, or 6.
* Female lactating patient, who will wean their children on starting treatment and ensure not to breastfeed after start treatment.
* Patients with an indication for SOF/DAC treatment for the treatment of chronic HCV.
* Patient is able and willing to sign the Informed Consent Form.
* Patient is able and willing to follow protocol requirements.

Exclusion Criteria:

* Need for co-treatment with ribavirin.
* HepBSAg positive test at screening.
* Treatment with rosuvastatin.
* Medicinal products that are potent P-glycoprotein (P-gp) and or CYP3A4 inducers in the intestine (rifampicin, rifabutin, St. John's wort [Hypericum perforatum], carbamazepine, phenobarbital and phenytoin).
* HIV co-infected patients using antiretroviral agents possibly interacting with SOF/DAC.
* Drugs associated with bradycardia including amiodarone.
* History of heart block.
* eGFR < 30 ml/min/1.73 m2.
* Compensated cirrhosis, based on historical data, evidence of decompensated cirrhosis by ascites, encephalopathy, or variceal hemorrhage and/or abnormal ALT/AST/INR/thrombocytes indicating cirrhosis.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion except for conditions related to HCV.
* Clinically relevant low hemoglobin concentration at screening.
* Pregnancy
* Refusal to use proper contraception during treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Lactating Women
Study Population: Lactating HCV infected female patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Plasma and milk concentrations of sofosbuvir | Time prior to first dose till 24 hours post first dose of sofosbuvir
  Determination of plasma and milk concentrations of sofosbuvir and its metabolite GS-331007 in plasma and milk of HCV infected lactating women.
Plasma and milk concentrations of daclatasvir | Time prior to first dose till 24 hours post first dose
  Determination of plasma and milk concentrations of daclatasvir in plasma and milk of HCV infected lactating women

CONTACTS AND LOCATIONS:
Overall Officials: Manal SE El-Sayed, M.D, Principal Investigator — Ain Shams University, Faculty of Medicine
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt